CLINICAL TRIAL: NCT01907906
Title: Inactivation of Whole Blood With Mirasol : Performance in Red Blood Cells in Healthy Volunteers
Brief Title: Inactivation of Whole Blood With Mirasol
Acronym: IMPROVEII
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Terumo BCTbio (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTS-0080; ERMS#12308001 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-06-20; First posted 2013-07-25 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Focus of Study: Radiolabel Recovery and Survival of RBCs
Keywords: Pathogen reduction technology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Mirasol-treated WB then untreated WB (Experimental): Screening Period (14 days); Treatment Period 1 (49 days): Donation of WB treated with Mirasol System for Whole Blood on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49); WB Donation Deferral Period (35-49 days); Treatment Period 2 (49 days): Donation of WB, UNTREATED on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49) Study Exit on Treatment Period 2, Day 49
  Interventions: Device: Mirasol System for Whole Blood
- Arm 2: Untreated WB then Mirasol-treated WB (Experimental): Screening Period (14 days); Treatment Period 1 (49 days): Donation of WB, UNTREATED on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49); WB Donation Deferral Period (35-49 days); Treatment Period 2 (49 days): Donation of WB treated with Mirasol System for Whole Blood on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49) Study Exit on Treatment Period 2, Day 49
  Interventions: Device: Mirasol System for Whole Blood

INTERVENTIONS:
Device: Mirasol System for Whole Blood — LR-pRBC units derived from WB will be treated with the Mirasol System. Treatment with the Mirasol System requires riboflavin to be mixed into the whole blood unit, which is then exposed to ultra violet (UV) light for a period of time; approximately an hour.
  Other Names: Pathogen Reduction Technology

SUMMARY:
The purpose of this study is to evaluate radiolabeled recovery and survival of autologous red blood cells (RBC), derived from Mirasol-treated fresh whole blood (WB), stored as leukoreduced packed RBC (LR-pRBC), and re-infused in healthy adult subjects

DETAILED DESCRIPTION:
This is a feasibility level study conducted to assess the recovery and survival of autologous, radiolabeled leukoreduced packed red blood cells (LR-pRBC) derived from fresh whole blood (WB) units that have been treated with the Mirasol System for Whole Blood (Mirasol System) and stored for 21 days at 1-6°C.1

ELIGIBILITY:
Inclusion Criteria:

* Eligible whole blood donor
* Age ≥ 18 years, of either sex
* Able to commit to the study follow-up schedule
* Subjects must have adequate bilateral antecubital venous access for WB collection and follow-up blood draws
* Negative screening test panel for infectious diseases
* Subjects of child-bearing potential (female or male) must agree to use effective contraceptive during the course of the study per site guidelines
* Subjects must agree to report adverse events (AEs) during the required reporting period
* Negative direct antiglobulin test (DAT) with subject's RBC
* Negative indirect antiglobulin test (IAT) with subject's serum

Inclusion for radiolabeled reinfusion of LR-pRBC on Day 21 (evaluated the day of, prior to, reinfusion):

* Maintenance of healthy status
* Negative direct antiglobulin test (DAT) with subject's RBC (fresh)
* Negative indirect antiglobulin test (IAT) with subject's serum (fresh) versus autologous stored LR-pRBC
* Negative serum or urine pregnancy test in females

Exclusion Criteria:

* Any serious medical illness and/or therapy, including: abnormal bleeding episodes, clotting or bleeding disorder, evidence of anemia, myocardial infarction, uncontrolled hypertension, heart disease, surgery with bleeding complications, epilepsy or any major surgery (with general or spinal anesthesia) within the last 6 months
* Pregnant or nursing females; For women of childbearing potential, negative serum or urine pregnancy tests at the time of WB donation and before the reinfusion are required
* Unable to give informed consent
* Participation currently, or within the last 12 months, in another investigational trial that would potentially interfere with the analysis of this investigation (e.g., pharmaceutical)
* Have received an accumulated radiation dose that would exclude them from the study according to the local radiation safety limits established by each institution
* Inability to comply with the protocol in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P Goodrich, PhD, Study Director — TerumoBCT Biotechnologies
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Puget Sound Blood Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Mirasol-treated Whole Blood (WB) Then Untreated WB: Screening Period (14 days); Treatment Period 1 (49 days): Donation of WB treated with Mirasol System for Whole Blood on Day 0, leuko-reduced packed red blood cells (LR-pRBCs) manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49); WB Donation Deferral Period (35-49 days); Treatment Period 2 (49 days): Donation of WB, UNTREATED on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49) Study Exit on Treatment Period 2, Day 49
Period: Overall Study
Arm/Group | Arm 1: Mirasol-treated Whole Blood (WB) Then Untreated WB | Arm 2: Untreated WB Then Mirasol-treated WB
Started | 16 | 13
Completed | 12 | 12
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: Adults ≥ 18 yrs; eligible WB donors with normal health status and vital signs by AABB criteria; negative infectious disease and direct/indirect antiglobulin test (DAT/IAAT), and did not meet any exclusion criteria.
Groups:
- Arm 2: Untreated WB Then Mirasol-treated WB: Screening Period (14 days); Treatment Period 1 (49 days): Donation of WB UNTREATED on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49); WB Donation Deferral Period (35-49 days); Treatment Period 2 (49 days): Donation of WB treated with Mirasol System for Whole Blood on Day 0, LR-pRBCs manufactured & stored 21 days, radiolabeled RBCs reinfused on Day 21 and samples collected over 28 days (Days 21-49)
- Total: Total of all reporting groups
Arm/Group | Arm 1: Mirasol-treated WB Then Untreated WB | Arm 2: Untreated WB Then Mirasol-treated WB | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 14 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 11 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell (RBC) 24-Hour Recovery
Description: To evaluate, as per FDA criteria, the 24-hour post transfusion RBC recovery in healthy adult subjects of leuko-reduced packed red blood cells (LR-pRBC) that have been derived from Mirasol-treated fresh WB units and stored at 1 to 6°C for 21 days.
  24-hour RBC Recovery is a measure of the % of RBCs that are still functioning 24 hours after they have been reinfused back into the donor following storage over 21 days.
Time Frame: 24 hours
Population: All subjects who signed an IC form (were enrolled), met eligibility criteria, had no intercurrent illness or notable signs/symptoms during the 24 hours prior to reinfusion, had no evidence of neoantigen formation on stored LR-pRBCs, and had at least 4 blood samples collected during the first 22 min, 30 sec post-infusion in each treatment period.
Measure: Mean (Standard Deviation); unit: % 24-hour RBC Recovery
Groups:
- Mirasol Treated: LR-pRBCs derived from Mirasol-treated WB
- Untreated Control: LR-pRBCs derived from untreated WB
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
% 24-hour RBC Recovery | 82.51 (3.914) | 91.70 (6.812)

2. Secondary Outcome: Red Blood Cell (RBC) Survival by Product
Description: Assessment of linear & exponential RBC survival and half-life (T50) over 28 days for RBCs derived from Mirasol-treated WB versus RBCs derived from untreated WB.
Time Frame: 28 days
Population: All subjects who signed informed consent,were eligible, had no intercurrent illness or notable signs/symptoms in 24 hrs prior to reinfusion, had no evidence of neoantigen formation on stored LR-pRBCs, and had ≥ 4 blood samples collected within the first 22 min 30 sec post-infusion in each treatment period.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Days
  Linear RBC Survival | 60.49 (5.574) | 81.57 (15.474)
  Linear T50 | 22.58 (4.328) | 35.83 (7.863)
  Exponential RBC Survival | 46.71 (5.630) | 67.81 (15.492)
  Exponential T50 | 22.63 (5.286) | 39.91 (10.485)

3. Secondary Outcome: Area Under the Curve (AUC) of Red Blood Cell (RBC) Survival
Description: Assessment of AUC of RBC survival over 28 days for RBCs derived from Mirasol-treated Whole Blood (WB) versus RBCs derived from untreated WB.
Time Frame: 28 days
Population: All subjects who signed an IC Form (were enrolled), met eligibility criteria, had no intercurrent illness or notable signs/symptoms during the 24 hours prior to reinfusion, had no evidence of neoantigen formation on stored LR-pRBCs, and had at least 4 blood samples collected within the first 22 min, 30 sec post-infusion in each treatment period.
Measure: Mean (Standard Deviation); unit: Days * Percent Recovery
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Days * Percent Recovery | 1715.2 (173.13) | 2055.2 (158.34)

4. Secondary Outcome: Spearman's Correlation Coefficients: 24-Hour Red Blood Cell (RBC) Recovery (%) With Hemolysis (%)
Description: Spearman's Correlation Coefficients comparing 24-Hour RBC Recovery (%) with Hemolysis (%) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 24 hours
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | -0.1779 | 0.4286

5. Secondary Outcome: Spearman's Correlation Coefficients: 24-Hour RBC Recovery (%) With Adenosine Triphosphate (ATP) (µmol/g Hgb)
Description: Spearman's Correlation Coefficients comparing 24-Hour RBC Recovery (%) with ATP (µmol/g Hgb) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 24 hours
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | 0.6107 | 0.4116

6. Secondary Outcome: Spearman's Correlation Coefficients: 24-Hour RBC Recovery (%) pCO2 (mmHg at 37° C)
Description: Spearman's Correlation Coefficients comparing 24-Hour RBC Recovery (%) with pCO2 (mmHg at 37° C) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 24 hours
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | 0.0383 | 0.0475

7. Secondary Outcome: Spearman's Correlation Coefficients: Linear T50 (Days) With Hemolysis (%)
Description: Spearman's Correlation Coefficients comparing Linear T50 (Days) with each of Hemolysis (%) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | -0.0592 | 0.0564

8. Secondary Outcome: Spearman's Correlation Coefficients: Linear T50 (Days) With Adenosine Triphosphate (ATP) (µmol/g Hgb)
Description: Spearman's Correlation Coefficients comparing Linear T50 (Days) with ATP (µmol/g Hgb) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | 0.2487 | 0.0261

9. Secondary Outcome: Spearman's Correlation Coefficients: Linear T50 (Days) With pCO2 (mmHg at 37° C)
Description: Spearman's Correlation Coefficients comparing Linear T50 (Days) with pCO2 (mmHg at 37° C) in packed Red Blood Cells (pRBCs) derived from Mirasol-treated whole blood (WB) versus pRBCs derived from untreated WB
Time Frame: 28 days
Population: as for outcome 3
Measure: Number; unit: Spearman's Correlation Coefficient
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Spearman's Correlation Coefficient | -0.0691 | -0.1065

10. Secondary Outcome: Neoantigenicity - Day 21 Direct Antigen Test (DAT)
Description: DAT testing of Red Blood Cells (RBCs) via Anti-immunoglobulin G (Anti-IgG) and Anti Complement Component 3 (Anti-C3) as derived from Mirasol-treated whole blood (WB) versus untreated WB conducted on Day 21 of both Treatment Periods 1 and 2. Number of positive results (indicating a new antigen formation) were recorded.
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test on Day 21 of both Treatment Periods 1 and 2
Measure: Number; unit: Positive results
Groups:
- Mirasol Treated: Leuko-Reduced packed Red Blood Cells (LR-pRBCs) derived from Mirasol-treated WB
- Untreated Control: Leuko-Reduced packed Red Blood Cells (LR-pRBCs) derived from untreated WB
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 23
Positive results | 0 | 0

11. Secondary Outcome: Neoantigenicity - Day 21 Indirect Antigen Test (IAT)
Description: Day 21 IAT testing of RBCs via LISS-15, Anti-IgG and C3 as derived from Mirasol-treated WB versus untreated WB. Number of positive results (indicating antibody formation to a new antigen) were recorded.
Time Frame: Day 21 of Treatment Periods 1 and 2
Population: as for outcome 10
Measure: Number; unit: Positive results
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 23
Positive results | 0 | 0

12. Secondary Outcome: Neoantigenicity - Day 42 Direct Antigen Test (DAT)
Description: DAT testing of RBCs via Anti-IgG and Anti-C3 as derived from Mirasol-treated WB versus untreated WB. Number of positive results (indicating a new antigen formation) were recorded.
Time Frame: Day 42 of Treatment Periods 1 and 2
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Number; unit: Positive results
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 23 | 24
Positive results | 0 | 0

13. Secondary Outcome: Neoantigenicity - Day 42 Indirect Antigen Test (IAT)
Description: IAT testing of RBCs via low ionic strength solution (LISS-15), Anti-IgG and C3 as derived from Mirasol-treated WB versus untreated WB. Number of positive results (indicating antibody formation to a new antigen) were recorded.
Time Frame: Day 42 of Treatment Periods 1 and 2
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test on Day 42 of both Treatment Periods 1 and 2.
Measure: Number; unit: Positive results
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
Positive results | 0 | 0

14. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Hematocrit (%)
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: % of volume
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
% of volume | 59.2 (2.83) | 61.0 (3.21)

15. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Hematocrit (%)
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: volume % of red blood cells
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 25 | 24
volume % of red blood cells | 58.3 (2.59) | 60.5 (2.65)

16. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - ATP
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: µmol/g Hgb
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
µmol/g Hgb | 4.659 (0.7372) | 4.544 (0.4275)

17. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - ATP
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: µmol/g Hgb
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
µmol/g Hgb | 4.416 (1.1313) | 5.403 (1.0111)

18. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - White Blood Cell (WBC) Count
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: 10E3 cells/µL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
10E3 cells/µL | 0.004 (0.0196) | 0.000 (0.0000)

19. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - White Blood Cell (WBC) Count
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: 10E3 cells/µL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 25 | 24
10E3 cells/µL | 0.004 (0.0200) | 0.021 (0.0833)

20. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Total Hemoglobin
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
g/dL | 19.4 (1.125) | 20.04 (1.222)

21. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Total Hemoglobin
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 25 | 24
g/dL | 19.26 (1.098) | 19.90 (1.097)

22. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - pH (at 37° C)
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: pH (at 37° C)
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
pH (at 37° C) | 6.8070 (0.03101) | 6.8253 (0.4117)

23. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - pH (at 37° C)
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 25 | 24
pH | 6.5537 (0.04776) | 6.5662 (0.04751)

24. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - pCO2 (mmHg at 37° C)
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: pCO2 (mmHg at 37° C)
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
pCO2 (mmHg at 37° C) | 59.16 (5.824) | 66.71 (6.607)

25. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - pCO2 (mmHg at 37° C)
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mmHg at 37° C
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 25 | 24
mmHg at 37° C | 93.09 (11.003) | 98.43 (10.438)

26. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Potassium
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
mEq/L | 2.17 (0.497) | 1.78 (0.465)

27. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Potassium
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
mEq/L | 65.50 (2.497) | 36.73 (3.749)

28. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Glucose
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
mg/dL | 560.3 (17.62) | 559.5 (45.88)

29. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Glucose
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
mg/dL | 408.5 (30.90) | 398.6 (33.84)

30. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Lactate
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 26 | 24
mmol/L | 2.39 (0.623) | 2.03 (0.561)

31. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Lactate
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
mmol/L | 17.54 (2.305) | 20.34 (3.092)

32. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Supernatant Hgb
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
mg/dL | 49.2 (16.66) | 47.1 (17.06)

33. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Supernatant Hgb
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
mg/dL | 99.6 (47.41) | 76.7 (34.60)

34. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - 2,3-diphosphoglycerate (DPG)
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: µmol/mL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
µmol/mL | 12.289 (2.1394) | 12.499 (3.7456)

35. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - 2,3-diphosphoglycerate (DPG)
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: µmol/mL
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
µmol/mL | 0.248 (0.2604) | 0.333 (0.4146)

36. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Hemolysis (%)
Time Frame: Day 0
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: % of volume
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
% of volume | 0.103 (0.0338) | 0.091 (0.0351)

37. Secondary Outcome: In Vitro Results From Leuko-Reduced Packed Red Blood Cells (LR-pRBCs) - Hemolysis (%)
Time Frame: Day 21
Population: All subjects who signed an IC Form (were enrolled), and had samples available for the requested test
Measure: Mean (Standard Deviation); unit: % of volume
Arm/Group | Mirasol Treated | Untreated Control
Number analyzed (Participants) | 24 | 24
% of volume | 0.215 (0.1001) | 0.150 (0.0606)

ADVERSE EVENTS:
Time Frame: All AEs collected from the first donation through the end of treatment period 2/study end - SAEs reported from time of 1st WB donation to study exit - TEAEs reported from time of LR-pRBC reinfusion on Day 21 to end of each treatment period
Description: Only Treatment Emergent AEs (TEAE) reported in final results. TEAEs = AEs that occurred following the Day 21 RBC reinfusion (24 total subj).
  SAE reporting: from 1st WB donation to study end (29 total subj). Per protocol, subjects were assessed for AEs at each study visit by site staff querying them on their general health since the previous visit
Arm/Group | Mirasol Treated | Untreated Control
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 11/24 | 11/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirasol Treated (N=24) | Untreated Control (N=24)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 5 | 5
Inflammation (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 5
Sinusitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less